CLINICAL TRIAL: NCT04195061
Title: Relative Sarcopenia and Cardiometabolic Risk in Young Adults With Obesity
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Melanie Schorr Haines, M.D, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2017P001495
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Overweight and Obesity; Insulin Resistance
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiopulmonary exercise testing
  Interventions: Procedure: Cardiopulmonary exercise test (CPET)

INTERVENTIONS:
Procedure: Cardiopulmonary exercise test (CPET) — CPET studies will be performed in the Cardiovascular Performance Program exercise lab at MGH. Subjects will undergo CPET on an upright cycle ergometer with continual measurement of metabolic gas exchange via a commercially available metabolic cart as well as heart rate and blood pressure. Exercise will proceed according to a maximal effort clinical protocol. Subjects will then undergo a standardized 30-min work load on the upright cycle ergometer based on the results of the maximal effort clinical protocol.

SUMMARY:
The goal of this research study is to learn more about the hormones that muscles make during exercise, and if those hormones are associated with type 2 diabetes risk in adults who are overweight or obese. Participants will undergo exercise testing on an upright bicycle, with blood samples taken for muscle hormones before and after exercise. The hypothesis is that adults with overweight/obesity and insulin resistance will have an impaired muscle hormone profile in response to exercise compared to adults with overweight/obesity who are not insulin resistant.

ELIGIBILITY:
Inclusion Criteria:

* Previously enrolled in protocol 2004P000013 or protocol 2012P002276, which had overweight or obesity as inclusion criteria
* Ability to walk up 3 flights of stairs and 3 city blocks (to ensure ability to complete exercise testing)

Exclusion Criteria:

* Unstable heart or lung disease
* Exercise >150 minutes/week
* Participation in college sports

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with overweight or obesity
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie S Haines, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin Sensitive: Homeostatic model assessment for insulin resistance (HOMA-IR) <1.9
- Insulin Resistant: Homeostatic model assessment for insulin resistance (HOMA-IR) >/=1.9
Period: Overall Study
Arm/Group | Insulin Sensitive | Insulin Resistant
Started | 19 | 9
Completed | 19 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Sensitive | Insulin Resistant | Total
Number analyzed (Participants) | 19 | 9 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (13.2) | 50.0 (12.0) | 53.4 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 11 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 15 | 8 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 16 | 5 | 21
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 9 | 28
Fasting serum myostatin [Mean (Standard Deviation); unit: ng/mL] | 9.84 (3.19) | 9.16 (2.34) | 9.62 (2.92)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 30.2 (4.0) | 40.8 (8.8) | 33.6 (7.7)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Serum Myostatin Levels From Pre- to 3 Hours Post-exercise
Description: Percent change in serum myostatin levels from pre- to 3 hours post-cardiopulmonary exercise test
Time Frame: Pre- to 3 hours post-exercise
Population: Four participants excluded from this analysis due to metformin use (n=2), testosterone use (n=1) or incomplete laboratory data (n=1).
Measure: Mean (Standard Deviation); unit: % change in serum myostatin
Groups:
- Insulin Sensitive: Homeostatic Model Assessment for Insulin Resistance < 1.9
- Insulin Resistant: Homeostatic Model Assessment for Insulin Resistance >/= 1.9
Arm/Group | Insulin Sensitive | Insulin Resistant
Number analyzed (Participants) | 17 | 7
% change in serum myostatin | -6.9 (41.8) | 8.5 (27.2)
Statistical Analysis 1: Comparison: Insulin Sensitive vs Insulin Resistant; Test type: Superiority; p = 0.303, t-test, 2 sided

2. Secondary Outcome: Percent Change in Serum Myostatin Levels From Pre- to 2 Hours Post-exercise
Description: Percent change in serum myostatin levels from pre- to 2 hours post-cardiopulmonary exercise test
Time Frame: Pre- to 2 hours post-exercise
Population: Four participants excluded from the analysis due to metformin use (n=2), testosterone use (n=1), or incomplete laboratory data (n=1).
Measure: Mean (Standard Deviation); unit: % change in serum myostatin
Arm/Group | Insulin Sensitive | Insulin Resistant
Number analyzed (Participants) | 17 | 7
% change in serum myostatin | -9.7 (39.4) | 21.7 (26.0)
Statistical Analysis 1: Comparison: Insulin Sensitive vs Insulin Resistant; Test type: Superiority; p = 0.035, t-test, 2 sided

3. Secondary Outcome: Percent Change in Serum Myostatin Levels From Immediately Post to 2 Hours Post-exercise
Description: Percent change in serum myostatin levels from immediately post to 2 hours post-cardiopulmonary exercise test
Time Frame: Immediately post to 2 hours post-exercise
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % change in serum myostatin
Arm/Group | Insulin Sensitive | Insulin Resistant
Number analyzed (Participants) | 17 | 7
% change in serum myostatin | -20.3 (36.0) | 13.5 (18.9)
Statistical Analysis 1: Comparison: Insulin Sensitive vs Insulin Resistant; Test type: Superiority; p = 0.007, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 week
Groups:
- Insulin Resistant: Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) >/= 1.9
Arm/Group | Insulin Sensitive | Insulin Resistant
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/9
Other Adverse Events (participants affected / at risk) | 0/19 | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Sensitive (N=19) | Insulin Resistant (N=9)
atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT04195061/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT04195061/SAP_001.pdf